CLINICAL TRIAL: NCT06949553
Title: OASIS PoST-Trial PAtient Registry (OASIS STAR)
Brief Title: An Observational Study to Learn More About Vasomotor Symptoms Burden and Treatment Patterns in Menopausal Women Before and After Participating in OASIS Studies
Acronym: OASIS STAR
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22884
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms (VMS) Associated With Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients who had participated in 1 of the 3 OASIS trials
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — No visits or examinations, laboratory tests or procedures are mandated or required for this study. Patients will be recruited through a registry if patients who had participated in previous OASIS trials. After this referral, the study is conducted entirely electronically.

SUMMARY:
This is an observational study to learn more about vasomotor symptoms (VSM) burden and treatment patterns in menopausal women before and after participating in OASIS studies.

In this study, data from women with VMS associated with menopause who took part in any of the three OASIS studies and were treated with elizanetant or a placebo, are collected and studied. In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

VMS associated with menopause is a condition in which women who have been through the menopause have hot flashes caused by hormonal changes. Menopause is the stage when a woman stops having menstrual cycles or periods.

No investigational products will be administered in this study. The participants in this study already received the standard of care (SOC) treatment for VMS before and after their participation in the study, as part of their regular care from their doctors. The SOC is the treatment that medical experts consider most appropriate currently.

OASIS is a set of clinical studies. In this study data will be collected from participants who took part in OASIS 1, 2 or 3 . These three studies assessed the safety and effects of elizanetant compared to a placebo for VMS associated with the menopause. Based on the results of these three studies, Bayer filed a New Drug Application for elizanetant.

To better understand the impact of elizanetant on VMS, more knowledge is needed about treatment patterns that were followed for VMS before and after the OASIS studies.

The main purpose of this study is to gather real-world data on participants' prescription trends, whether they continued or stopped taking treatments, and healthcare resource utilization, before and after their participation.

This study will include participants from OASIS 1,2 or 3 from the United States of America, who have agreed to be contacted to share information regarding their treatment. This study will have 2 parts:

Part A - researchers will invite participants to complete an online survey about the treatments given in the year before starting the OASIS study.

Part B - researchers will use tokens (an anonymized number to ensure participants' privacy) to learn about the treatments given to them 6 months after the completion of the OASIS study through their anonymized medical records.

Researchers will collect the following information:

Part A:

* the prescription and over-the-counter medicines used by the participants for VMS in the year before the OASIS start
* whether they continued or stopped taking them, and
* the reason for doing so

Part B:

* the prescription medicines used by the participants for VMS in 6 months after the OASIS ended
* whether they continued or stopped taking them

For Part A the data will be collected from the participant survey between March 2025 and June 2025, and for Part B the data will be collected using participants' medical records between April 2025 to May 2025.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the US who participated in one of the three OASIS trials for patients with moderate-to-severe VMS related to menopause.
* Patients who confirmed interest in being contacted for further study communication
* Patients who consent to be included in the registry, complete the pre-OASIS trial survey, and agree to be tokenized so that their anonymized real-world data can be accessed

Exclusion Criteria:

* None

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women experiencing menopause assigned female at birth
Study Population: Females from 40 to 65 years, naturally or surgically postmenopausal, who had experienced 50 or more moderate to severe VMS over 7 days during screening
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Prescription medication(s) used to treat VMS (Vasomotor symptoms) related to menopause | Survey will remain open from Day 1 up to 12 weeks after Day 1.
  Measured using a one time Web-based survey. Survey collects retrospective information from 12 months before the FPFV (range from 27AUG2021 to 29OCT2021) of one of the three OASIS studies.
Use of OTC (over the counter) medicines to treat moderate-to-severe VMS related to menopause | Survey will remain open from Day 1 up to 12 weeks after Day 1.
  Measured using a one time Web-based survey. Survey collects retrospective information from 12 months before the FPFV (range from 27AUG2021 to 29OCT2021) of one of the three OASIS studies.
Use of non-pharmaceutical therapies to treat moderate-to-severe VMS related to menopause | Survey will remain open from Day 1 up to 12 weeks after Day 1.
  Measured using a one time Web-based survey. Survey collects retrospective information from 12 months before the FPFV (range from 27AUG2021 to 29OCT2021) of one of the three OASIS studies.
Adherence to prescribed and OTC medication and reasons for non-adherence | Survey will remain open from Day 1 up to 12 weeks after Day 1.
  Measured using a one time Web-based survey. Survey collects retrospective information from 12 months before the FPFV (range from 27AUG2021 to 29OCT2021) of one of the three OASIS studies.
Discontinuation of prescribed and OTC medication and reasons for discontinuation | Survey will remain open from Day 1 up to 12 weeks after Day 1.
  Measured using a one time Web-based survey. Survey collects retrospective information from 12 months before the FPFV (27AUG2021-29OCT2021) of one of the three OASIS studies.
Prescription medications used to treat VMS related to menopause | Retrospective analysis from12 months before the FPFV (range from 27AUG2021 to 29OCT2021) and 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)
Adherence to prescribed medication | Retrospective analysis from12 months before the FPFV (range from 27AUG2021 to 29OCT2021) and 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)
Discontinuation of prescribed medication | Retrospective analysis from12 months before the FPFV (range from 27AUG2021 to 29OCT2021) and 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)

SECONDARY OUTCOMES:
Treatment pattern for VMS medications in the 12-month period prior to initiation of the OASIS trial and the month post-OASIS trial period | Retrospective analysis from12 months before the FPFV (range from 27AUG2021 to 29OCT2021) and 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)
Time from OASIS trial completion and 4-week follow-up to start of each VMS treatment | Retrospective analysis after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies
  Collected from external linked data source(s)
Frequency of outpatient office visits by specialty of healthcare provider (HCP) | Retrospective analysis from 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)
The 5 most common reasons for outpatient visits | Retrospective analysis from 6 months after LPLV (range from 10OCT2023 to 12FEB2024) of one of the three OASIS studies.
  Collected from external linked data source(s)

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer US, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.